CLINICAL TRIAL: NCT03962517
Title: Effect of GEMS-H on Locomotor Function in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Electronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-04-063
Record Dates: First submitted 2019-05-20; First posted 2019-05-24 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Adults; Middle Age; Aged; Aged, 80 and Over

STUDY DESIGN:
Intervention Model Description: Training in the GEMS-H group consists of 15 minutes task-specific training and 30 minutes functional gait training on varied environments with device, whereas training in the control group consists of 15 minutes task-specific training and 30 minutes functional gait training on varied environments without device.
Who Masked: Outcomes Assessor
Masking Description: A blinded research physical therapist will test the outcome measure at baseline, mid testing after 9th session of training, at post testing after 18th session of training, at 1 month follow up testing after 18th session of training and at 3 months follow up testing after 18th session of training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training with GEMS-H (Experimental): Participants will participate in 18 sessions of training + 5 sessions of testing for up to 3 month.
  Training consists of 15 minutes task-specific training and 30 minutes functional gait training on varied environments with the device.
  Interventions: Device: with Gait Enhancing and Motivating System-Hip (GEMS-H)
- Training without GEMS-H (Active Comparator): Participants will participate in 18 sessions of training + 5 sessions of testing for up to 3 month.
  Training consists of 15 minutes task-specific training and 30 minutes functional gait training on varied environments without the device.
  Interventions: Other: without Gait Enhancing and Motivating System-Hip (GEMS-H)

INTERVENTIONS:
Device: with Gait Enhancing and Motivating System-Hip (GEMS-H) — The intensity of training: between 12 and 16 in borg's rating of perceived exertion scale.
  Assessments consist of gait function, cardiopulmonary metabolic energy cost, physical performance, balance, physical level, pain, fall efficacy, depression, quality of life and activities of daily living.
  Arms: Training with GEMS-H
Other: without Gait Enhancing and Motivating System-Hip (GEMS-H) — The intensity of training: between 12 and 16 in borg's rating of perceived exertion scale.
  Arms: Training without GEMS-H

SUMMARY:
The purpose of this study is to investigate the effect of training with the Gait Enhancing and Motivating System-Hip (GEMS-H) vs. training without the GEMS-H on locomotor function in adults. The investigator hypothesizes that long-term GEMS-H use would improve locomotor function. Specifically, individuals in the GEMS-H group will show faster gait speed compared to those in the control group.

DETAILED DESCRIPTION:
The GEMS-H is a hip-type assist device developed by Samsung Electronics. The GEMS-H is worn around the waist and fastened at the waist and thighs by a set of belts with velcro to assist motion at the hip joints. The device weighs 2.1kg, and has 2 brushless direct current motors running on a rechargeable lithium ion battery. The normal operation time for the device is 2 hours. It is controlled through a custom built application on a hand held tablet.

The purpose of this study is to investigate the effect of training with the Gait Enhancing and Motivating System-Hip (GEMS-H) vs. training without the GEMS-H on locomotor function in adults. The investigator hypothesizes that long-term GEMS-H use would improve locomotor function. Specifically, individuals in the GEMS-H group will show faster gait speed compared to those in the control group.

Participants will be scheduled for 18 sessions of training (randomly placed either in GEMS-H training group or traditional training group without the GEM-H) plus 5 sessions of testing (pre-training, mid-test after the 9 sessions of training, post-training, 1 month follow-up and 3 month follow-up after the 18 sessions training completed).

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 - 84 years
* No history of central nervous system related disease

Exclusion Criteria:

* Difficulty in walking due to conditions such as poor vision or fractures
* Height is less than 140cm or more than 185cm.
* Body mass index (BMI) greater than 35.
* Difficulty understanding and participating in the study such as those with cognitive problems or dementia.
* Subject who is at risk of falling during walking due to severe dizziness

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Change in 10 Meter Walk Test-Self Selected Velocity (sec) from Baseline to Post-Training Assessment | Baseline Assessment, Post Training Assessment (6 weeks)
  Measure of self-selected walking speeds by measuring the time it takes a participant to walk 10 meters. The test is performed using a "flying start," the participant walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Change in 10 Meter Walk Test-Fast Velocity (sec) from Baseline | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  Measure of fast walking speeds by measuring the time it takes a participant to walk 10 meters. The test is performed using a "flying start," the participant walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance as fast as you can safely when I say go."
Change in 10 Meter Walk Test-Self Selected Velocity (sec) from Baseline to Other Assessment Time Points | Baseline Assessment, Mid Training Assessment (3 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  Measure of self-selected walking speeds by measuring the time it takes a participant to walk 10 meters. The test is performed using a "flying start," the participant walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."
Functional Gait Assessment (FGA) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The FGA is used to assess postural stability during walking and assesses a participant's ability to perform multiple motor tasks while walking. The tool is a modification of the 8-item Dynamic Gait Index, developed to improve reliability and reduce ceiling effect. Scores of 22/30 on the FGA is effective in predicting falls.
Short Physical Performance Battery (SPPB) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The SPPB is an assessment tool for evaluation of lower extremity function.
Functional Reach Test (FRT) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The FRT assesses a participant's stability by measuring the maximum distance the participant can reach forward while standing in a fixed position.
Four Square Step Test (FSST) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The FSST is used to assess dynamic stability and the ability of the participant to step over low objects forward, sideways, and backward
Five times Sit to Stand (5xSST) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The 5XSST is used to assess functional lower extremity strength, transitional movements, balance, and fall risk. The instructions are: "Please stand up straight as quickly as you can 5 times, without stopping in between. Keep your arms folded across your chest. I'll be timing you with a stopwatch. Ready, begin."
Berg Balance Scale (BBS) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The BBS is a 14-item objective measure that assesses static balance and fall risk.
Timed Up and Go test (TUG) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The TUG is a simple test used to assess a participant's mobility and requires both static and dynamic balance. TUG uses the time that a participant takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the participant is expected to wear their regular footwear and use any mobility aids that they would normally require.
Wearable activity tracker (Measurement: Step count, Calorie consumption, and Heart rate) | Up to Post Training Assessment (Up to 6 weeks)
  Each participant is given an activity monitor band and instructed to wear it on the wrist during waking hours until completion of the training program (between Visit 2 and Visit 21).
EuroQol 5 Dimensions (EQ-5D) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)]
  The EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the participant's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are.
Korean-Modified Barthel Index (K-MBI) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The K-MBI is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
Fall Efficacy Scale-Korean (FES-K) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The FES-K is the measures of "fear of falling" or, more properly, "concerns about falling", which are suitable for use in research and clinical practice.
Visual Analogue Scale (VAS) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The VAS is a pain rating scale. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale; "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Geriatric Depression Scale-a short version (GDS-SF) | Baseline Assessment, Mid Training Assessment (3 weeks), Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The GDS is a 15-item self-report assessment used to identify depression in the elderly. A score of 0 to 5 is normal. A score greater than 5 suggests depression.
Change in Muscle Strength from Baseline | Baseline Assessment, Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  The maximal isometric strength of the 12 muscles in lower extremity will be measured with 12 channels surface electromyography (NORAXON™, USA).
Change in Muscle Activation Pattern and Effort (%MVC) during Gait from Baseline | Baseline Assessment, Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  All participants perform over-ground walking to assess the change of muscle activation pattern and effort (%MVC) using 12channels surface EMG
Change in Gait Function from Baseline | Baseline Assessment, Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  All participants perform over-ground walking to assess the change of kinematic (lower extremity joint angles), kinetics (lower extremity joint moments) and ground reaction force using motion analysis (Kestrel Digital RealTime System, Motion Analysis Corporation, USA) and force plate ( TF-4060-B, Tec Gihan Co., Ltd. Japan), respectively.
Change in Cardiopulmonary Metabolic Energy Consumption from Baseline | Baseline Assessment, Post Training Assessment (6 weeks), 1 month Post Training Assessment (1 month Follow-up), 3 month Post Training Assessment (3 month Follow-up)
  All participants perform treadmill 6 minute walk test (6MWT) to assess the change of metabolic energy expenditure using a portable cardiopulmonary metabolic system (Cosmed K4b², Rome, Italy).

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea